CLINICAL TRIAL: NCT00834548
Title: Whole-Body MRA at 3T - A Comparison Between Two Different Scan Protocols
Status: Completed | Type: Observational
Sponsor: Copenhagen University Hospital at Herlev (Other)
Collaborators: Rigshospitalet, Denmark (Other)
Responsible Party: Yousef Nielsen MD, Copenhagen University Hospital Herlev
Other Study IDs: Herlev WB-MRA 5
Record Dates: First submitted 2008-08-26; First posted 2009-02-03 (Estimated); Last update posted 2009-02-03 (Estimated); Status verified 2009-02

CONDITIONS: Atherosclerosis; Intermittent Claudication
Keywords: Magnetic resonance; whole body; angiography; hybrid protocol; MRI
MeSH Terms: conditions — Atherosclerosis; Intermittent Claudication

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 1: WB-MRA standard protocol
  Interventions: Procedure: Whole body magnetic resonance angiography (WB-MRA)
- 2: WB-MRA hybrid protocol
  Interventions: Procedure: Whole body magnetic resonance angiography (WB-MRA)

INTERVENTIONS:
Procedure: Whole body magnetic resonance angiography (WB-MRA) — WB-MRA will be performed once in each patient.

SUMMARY:
To compare to different approaches in whole-body magnetic resonance angiography of patients suffering peripheral arterial disease.

Our hypothesis is that use of a new protocol improves the diagnostic quality of the WB-MRA procedure.

DETAILED DESCRIPTION:
Patients suffering peripheral arterial disease must undergo imaging procedures before endovascular or surgical procedures.

WB-MRA is an imaging procedure that can visualise the arterial system. WB-MRA can be performed in different manners. On option is to start the scan in the head region and continue down the body to the feet (standard protocol). Another option is to use a hybrid protocol that first examines the head and lower leg followed by examination of the pelvic and upper leg region.

A comparison between the standard and hybrid protocols has not been performed in a 3T high magnetic field system, therefore we will perform such a study.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic lower extremity ischemia (claudication, ischemic wounds)
* Referred to digital subtraction angiography (DSA)

Exclusion Criteria:

* Renal insufficiency (GFR < 30 ml/min)
* Contra-indications for MRI-examination (claustrophobia, metal-implants, pacemaker)
* Dementia
* Pregnancy/lactation
* Allergy to gadolinium based MRI contrast agents
* Acute disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with peripheral arterial disease
Enrollment: 26 (Estimated)
Dates: Start 2008-06; Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Diagnostic quality of WB-MRA

SECONDARY OUTCOMES:
Signal to noise ratio
Contrast to noise ratio

CONTACTS AND LOCATIONS:
Overall Officials: Yousef W Nielsen, MD, Principal Investigator — Copenhagen University Hospital at Herlev
Locations (1):
- Copenhagen University Hospital Herlev, Herlev Copenhagen, Denmark